CLINICAL TRIAL: NCT04206540
Title: Effect of Electrical Stimulation of the Auricular Branch of the Vagus Nerve (ABVN) on Cervical Vagus Nerve Compound Nerve Action Potentials(CNAPs)
Brief Title: Effect of Stimulation on the Vagus Nerve
Acronym: ABVN1
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Purdue University (Other)
Responsible Party: Principal Investigator, Thomas V. Nowak, Clinical Professor and Principal Investigator, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1809683671; 1809683671 (Other: IRB)
Record Dates: First submitted 2019-12-18; First posted 2019-12-20 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Healthy Subjects (Experimental): Healthy volunteers aged 18-80 years old who will undergo vagus nerve stimulation.
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation; Procedure: Vagal Stimulation

INTERVENTIONS:
Device: Transcutaneous Auricular Vagus Nerve Stimulation — Electrical stimulation of the vagus nerve around the external ear using a transcutaneous device. Electrical current will be increased in intensity based on subject feedback of a scale 0-10.
  Electrical stimulation will be delivered for 2 minutes once the subject reports the maximum comfortable intensity.
  Other Names: ML1101 Stimulus Isolator
Procedure: Vagal Stimulation — Subjects will be asked to do the following in order to stimulate the vagus nerve:
  * Cough 6 to 8 forceful coughs
  * Have an ice cold wash cloth placed on their face for 10 seconds.
  * Carotid massage
  * Gagging: a tongue depressor is briefly inserted into the back of the mouth touching the bag of the throat.
  * Valsalva maneuver: Subjects will be asked to bear down as if having a bowel movement. They will be asked to blow through a mouthpiece that is hooked to a device that measures how hard they are blowing. Alternatively, we can have them blow through the barrel of a 10 ml syringe for 15-20 seconds.
  * Eating: Subjects will be asked to drink water and/or Ensure that has 220 calories after fasting overnight.
  Other Names: Vagal Maneuvers

SUMMARY:
The vagus nerve is a largely-internal nerve that controls many bodily functions, including stomach function. Investigators hope that electrically stimulating the nerve around the external ear will also stimulate the internal vagus nerve. If it does, then investigators hope that this will help the treatment of patients with nausea and vomiting and disordered stomach function.

Investigators also hope to be able to measure the activity of the vagus nerve when it is stimulated in other ways. This could help investigators learn more about studying this nerve in the future.

DETAILED DESCRIPTION:
Only healthy volunteer subjects will be recruited and studied for this project. Volunteer subjects will undergo transcutaneous stimulation of the auricular branch of the vagus nerve (ABVN) to determine whether this modality will also produce cervical vagus nerve compound action potentials. Ear Stimulation Group

Another part of the study is to measure the vagal response to maneuvers which are known to stimulate the vagus nerve. The implementation of these vagal maneuvers will allow comparison of ABVN stimulation to traditional methods of vagal stimulation.- Vagal Maneuver Group

EAR STIMULATION GROUP:

This is a onetime visit only that involves baseline and test procedures.

Two MRI compatible electrodes will be placed in the auricle of the left ear, fixed by a plastic armature that wraps around the ear. The leads from the electrodes are connected to a stimulator.

A pneumatic belt may be placed around the lower thorax. Pneumatic tubes connect this belt to a pressure transducer that in turn sends signal to a laptop-controlled device that acquires the signals.

Two ECG electrodes are placed on both sides of the neck overlying the area near the carotid artery where the vagus nerve is superficial. This is to measure the vagal action potentials in the neck. Two ECG electrodes are placed one on each arm and one on the chest for measurement of the electrocardiogram (ECG ). Three ECG electrodes are placed on the abdomen in a line parallel to the longitudinal axis of the stomach to record the electrogastrogram (EGG). Electrical stimulation of the electrodes placed in the ear is provided by a current-constant stimulator. The stimuli consist of rectangular pulses with 450 µs pulse width, delivered at 30 Hz, and pulse train duration of 0.5 seconds. Stimulation is gated, with 0.5-second delay, after peak inhalation (i.e., during exhalation) or after peak exhalation (i.e., during inhalation).

Baseline procedure:

During the baseline recording the stimulating electrodes are placed in the auricle of the subject but no current is delivered. Cervical neck electrodes are placed over the right and left vagus nerve to record any electrical activity that might occur during the baseline period. Baseline ECG and EGG recordings are also performed during this interval.

Test procedure:

Stimuli consisting of rectangular pulses with 450 µs pulse width, delivered at 30 Hz, and pulse train duration of 0.5 seconds are then delivered to the subject. Current intensity is set to achieve moderate to strong (but not painful) sensation, and pulse frequency/duration is set following pilot testing to achieve a subjectively comfortable stimulus sensation. This level of current stimulation is designated "100 per cent." The current is then reduced to 10 per cent and ABVN is continued for 60 seconds. The current amplitude is then increased again by 10 per cent and ABVN is applied again for 60 seconds. This sequence is repeated until the "100 percent" level is reached. These stimuli are delivered during expiratory phase of respiration as investigations have shown this to be most effective in producing vagal stimulation (8).

Once the target stimulus intensity has been achieved, stimuli are delivered during the expiratory phase for a total of two minutes. Stimuli are then delivered at 50% and 25% of the original amplitude for 2 minutes, respectively.

ECG and EGG recordings are continued during auricular branch vagal nerve stimulation.

VAGAL MANEUVER GROUP:

Healthy volunteers will be recruited initially to see the effect of these maneuvers on the vagal activity.

A total of 30 healthy volunteers will be recruited. At the beginning of the study, a baseline recording of 10 minutes will be made following which the maneuvers will be conducted. Cervical neck electrodes are placed over the right and left vagus nerve to record any electrical activity that might occur during the baseline period. Baseline ECG and EGG recordings are also performed during this interval by placing the electrodes over the chest and over the stomach area for ECG and EGG recordings.

After 10 seconds of each maneuver, another 8 minutes of recording will be made before doing the next maneuver.

For the eating maneuver there is no time restriction and the subject will drink it as per their capacity. After drinking the Ensure, a 20 minute recording will be made.

Investigators will include the following maneuvers:

Cough; Each subject will be asked to generate approximately 6 to 8 forceful and sustained coughs over 5 to 10 seconds.

Cold stimulus to face: This technique involves submerging a patient's face in ice cold water. We propose to place an ice pack or a washcloth soaked in ice water on each subject's face for about 10 seconds. This creates a physiological response to a person being submerged in cold water (Diver's Reflex) Carotid Massage: This technique is performed with the subject's neck in an extended position, the head turned away from the side being massaged. Only one side is massaged at a time. Pressure is applied underneath the angle of the jaw in a gentle circular motion for about 10 seconds. The subject is monitored throughout.

Gagging: A tongue depressor is briefly inserted into the subject's mouth touching the back of the throat, which causes the person to reflexively gag. The gag reflex stimulates the Vagus nerve.

Valsalva maneuver: The subject is instructed to bear down as if they were having a bowel movement. The subject is asked to blow through a mouthpiece that is hooked to a device used in clinical spirometry until the pressure reaches 10mmHg. Alternatively, we can have the subject blow through the barrel of a 10 ml syringe for 15-20 seconds. This maneuver increases intrathoracic pressure and stimulates the Vagus nerve.

Eating: Subjects will be asked to drink Ensure Original that has 220 calories after fasting overnight to see that effect on vagal activity during eating.

All the maneuvers described above will be conducted for duration of 10 seconds each except wherever stated otherwise and the recordings will be made for duration of 8 minutes after each maneuver. If it is not possible to all the maneuvers in one visit then they will be conducted over two visits. Sometimes not all maneuvers will be conducted and this will depend on the discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers
2. Aged 18-80 years
3. Willing to have electrodes placed in the external ear (ABVN arm)
4. Willing to perform vagal activity maneuver ( Vagal arm)

Exclusion Criteria:

1. Unable to provide consent
2. Having gastric motility issues as determined by the PI or Sub I
3. Taking medications affecting gastric motility
4. Pregnant females
5. Prisoners

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-07-22 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Amplitude of the Vagus nerve with ABVN | 3 years
  measure the amplitude of vagal nerve compound action potentials in healthy volunteers with skin electrodes over right and left vagus nerve during ABVN stimulation
Amplitude of Vagus Nerve with Vagal Maneuvers | 3 years
  measure the amplitude of vagal nerve compound action potentials in healthy volunteers with skin electrodes over right and left vagus nerve during Vagal Maneuvers.

SECONDARY OUTCOMES:
EGG and ABVN | 3 years
  Measure changes in the amplitude of the surface electrogastrogram(EGG) during ABVN
EGG and Vagal maneuver | 3 years
  Measure changes in the amplitude of the surface electrogastrogram(EGG) during Vagal Maneuver

CONTACTS AND LOCATIONS:
Overall Officials: Thomas V Nowak, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Hosptial, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No